CLINICAL TRIAL: NCT05180487
Title: Rural Families Affected by Opioid Use: An Online Parenting Intervention; and Supplement to Prevention Research Center: Parenting Among Women Who Are Opioid Users, Project 2
Brief Title: Parenting Young Children Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10212019.029; P50DA048756 (NIH); P50DA048756-01S1 (NIH)
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Parenting; Parent-Child Relations; Opioid Misuse; Opioid Use Disorder; Stress; Depression; Parenting Self-efficacy
MeSH Terms: conditions — Opioid-Related Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Families will be assigned to treatment vs. wait-list control. The investigators will assess families at baseline and at 3-, 6-, and 12-month follow-ups. Families in the treatment condition will receive the intervention between baseline and the 3-month follow-up. The control group will receive the intervention following the 12-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCU Online + Coach (Experimental): Parents in this arm will receive access to the FCU Online website and telehealth coaching/ support provided by a trained mental health provider. The FCU Online website includes a brief 5-minute assessment, feedback on parents' responses, and online tools to support parenting in areas that were identified as challenges by the assessment. These tools include animated videos, parenting tips, and interactives to help practice parenting skills. Telehealth coaching will focus on Wellness and Self-Care, Parenting and Substance Use, Positive Parenting, Proactive Parenting, and Supervision and Limit Setting.
  Interventions: Behavioral: Family Check-Up
- Waitlist Control (No Intervention): Parents in this arm will initially serve as the control group but will receive access to the FCU Online website after completing four waves of data collection (baseline, 3-mo, 6-mo, and 12-mo follow-up).

INTERVENTIONS:
Behavioral: Family Check-Up — This intervention includes access to the Family Check-Up Online website and telehealth coaching provided by trained mental health providers. A minimum of 5 coaching sessions will be provided.
  Arms: FCU Online + Coach

SUMMARY:
Opioid use is rising at unprecedented levels and has reached epidemic proportions in some areas of the country, particularly rural areas. Although research on the detrimental effects of opioid use on parenting and children is relatively new, it is clear that parents with opioid use struggle with a variety of parenting skills, especially contingent responsivity and warmth. As such, to have long-term sustained effects on preventing Opioid Use Disorder (OUD) in parents and to help prevent substance use and related problem behaviors in the next generation, it is critical to prevent opioid use, opioid misuse, and OUD in new parents, in tandem with providing support for parenting skills.

The Family Check-Up Online (FCU Online) focuses on supporting parents by increasing parenting self-efficacy, stress management skills, self-regulation skills, and sleep routines, which are hypothesized to lead to the prevention of opioid misuse and OUD as well as improve mental health and increase responsive parenting. The FCU Online is based on the Family Check-Up, which has been tested in more than 25 years of research, across multiple settings, and is an evidence-based program for reducing high-risk behavior, enhancing parenting skills, and preventing substance use through emerging adulthood. It is named in NIDA's "Principles of Substance Use Prevention for Early Childhood" as one of only three effective selective prevention programs for substance abuse among families with young children. The FCU has also been endorsed as an evidence-based practice by the Maternal Infant and Early Childhood Home Visiting Program (MIECHV), and has been listed as a promising program by the Blueprints for Healthy Youth Development since 2013.

The current project aims to address barriers of access to prevention services by delivering the FCU in a telehealth model using the FCU Online. In this research study the investigators will:

1. Work with community stakeholders in rural Oregon to expand the FCU Online to target early childhood (ages 18 months-5 years) and mothers with opioid misuse and addiction. Guided by focus group feedback, the FCU Online will be adapted to target parenting skills relevant to mothers with opioid misuse, including positive parenting, parent-child relationship building, executive functioning to help manage stress and depression, and negative parenting. A 2-month feasibility study (n=10) will test the adapted version of the FCU Online and help investigators refine intervention procedures and usability, recruitment steps, and assessment delivery.
2. Examine the efficacy of the FCU Online for rural families with opioid or other substance misuse. 400 parents with preschool children ages 18 months to 5 years and who have been identified with substance misuse, opioid misuse, or addiction will be randomly assigned to receive the FCU Online or services as usual and followed for one year. A telehealth model will be used for intervention delivery that includes targeted coaching and support. The investigators predicted that parents assigned to the FCU Online intervention will (a) show improvements in parenting skills linked to improvements in child behavior and long-term risk for subsequent substance abuse, and (b) show improvements in self-regulation and executive functioning (inhibitory control, attention shifting), which will mediate intervention effects. The investigators will also examine moderators, including neonatal abstinence syndrome/neonatal opioid withdrawal syndrome, and model intervention effects over time.
3. Examine factors related to successful uptake and implementation. To facilitate dissemination on a national scale, investigators will assess the feasibility of the FCU as an Internet-delivered intervention in rural communities with high levels of opioid use, including the extent to which participants engaged in the intervention, completed the program, and were satisfied with the program. Investigators will also assess feasibility, usage, fidelity, and uptake through engagement data collected via the online web portal. The investigators will develop materials and briefings for community agencies that will increase knowledge dissemination and, ultimately, reach a greater number of families throughout the United States who need information and services for parenting support in the context of opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* Must be a parent or legal guardian of a child between the ages of 18 months and 5 years old that lives in the parent's home at least 50% of time;
* Must have a smart phone with text messaging capability and access to email;
* Must be willing to complete phone interviews and use a telehealth program that focuses on strengthening parenting;
* Must respond 'yes' to binge drinking and/or recreational drug use in the last year, lifetime use of prescription opioids, or depressed mood in the last two weeks.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stormshak, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon Prevention Science Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 947 parents inquired about study participation. Some were excluded due to being unresponsive to outreach (n=289), inquiring after recruitment was closed (n=12), not meeting inclusion criteria (n=244), or declining to participate (n=20). 382 parents qualified to participate, and 356 completed the consent process and baseline data collection. Parents who returned baseline surveys (n=356) were randomly assigned to one of two conditions.
Period: Baseline
Arm/Group | FCU Online + Coach | Waitlist Control
Started | 180 | 176
Completed | 180 | 176
Not Completed | 0 | 0
Period: 3-month Follow-up
Arm/Group | FCU Online + Coach | Waitlist Control
Started | 169 | 169
Completed | 169 | 169
Not Completed | 0 | 0
Period: 6-month Follow-up
Arm/Group | FCU Online + Coach | Waitlist Control
Started | 163 | 165
Completed | 163 | 165
Not Completed | 0 | 0
Period: 12-month Follow-up
Arm/Group | FCU Online + Coach | Waitlist Control
Started | 165 | 162
Completed | 165 | 162
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FCU Online + Coach | Waitlist Control | Total
Number analyzed (Participants) | 180 | 176 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: N=355 for this question, rather than N=356, because data is missing for one participant in the FCU Online + Coach condition.
  years
    number analyzed (Participants) | 179 | 176 | 355
    (all) | 33.77 (5.64) | 33.59 (6.30) | 33.68 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: N=354 for this question, rather than N=356, because two participants in the waitlist control condition chose not to respond to this demographic question.
  Participants
    number analyzed (Participants) | 180 | 174 | 354
    Female | 169 | 161 | 330
    Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 38 | 75
  Not Hispanic or Latino | 140 | 135 | 275
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 1 | 5 | 6
  White | 136 | 134 | 270
  More than one race | 33 | 30 | 63
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 180 | 176 | 356

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parenting Skills: Supporting Positive Behavior
Description: Parents' skill in supporting positive behavior was measured with the "supporting positive behavior" subscale of the Parenting Young Children Questionnaire (PARYC). Scores could range from 7-49; a higher score indicates greater skill in supporting positive behavior.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning surveys at follow-up waves).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 176 | 171
score on a scale
  baseline | 37.35 (5.61) | 37.43 (6.54)
  3-month follow up: number analyzed (Participants) | 160 | 159
  3-month follow up | 38.51 (5.33) | 37.49 (6.49)
  6-month follow up: number analyzed (Participants) | 157 | 156
  6-month follow up | 39.01 (5.59) | 37.13 (6.06)
  12-month follow up: number analyzed (Participants) | 151 | 151
  12-month follow up | 39.30 (5.74) | 37.71 (6.37)

2. Primary Outcome: Change From Baseline in Parenting Skills: Setting Limits
Description: Parents' skill in setting limits was measured with the "setting limits" subscale of the Parenting Young Children Questionnaire (PARYC). Scores could range from 7-49; a higher score indicates greater skill in setting limits.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 177 | 171
score on a scale
  baseline | 35.40 (6.13) | 35.04 (6.70)
  3-month follow up: number analyzed (Participants) | 160 | 161
  3-month follow up | 38.72 (5.60) | 36.35 (5.84)
  6-month follow up: number analyzed (Participants) | 158 | 159
  6-month follow up | 38.68 (7.07) | 36.43 (6.52)
  12-month follow up: number analyzed (Participants) | 152 | 151
  12-month follow up | 39.34 (6.51) | 36.75 (6.63)

3. Primary Outcome: Change From Baseline in Parenting Skills: Proactive Parenting
Description: Parents' skill in proactive parenting was measured with the "proactive parenting" subscale of the Parenting Young Children Questionnaire (PARYC). Scores could range from 7-49; a higher score indicates greater skill in proactive parenting.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 177 | 171
score on a scale
  baseline | 36.45 (6.95) | 35.49 (7.64)
  3-month follow up: number analyzed (Participants) | 161 | 160
  3-month follow up | 40.04 (5.54) | 36.68 (6.82)
  6-month follow up: number analyzed (Participants) | 158 | 159
  6-month follow up | 40.04 (6.60) | 37.57 (7.24)
  12-month follow up: number analyzed (Participants) | 153 | 152
  12-month follow up | 39.84 (6.76) | 37.69 (6.95)

4. Primary Outcome: Change From Baseline in Parenting Confidence
Description: Parents' confidence in their parenting skills was measured with the Behavioral Self-Efficacy subscale (PAREFF) of the Parenting Tasks Checklist. Scores could range from 1-5; a higher score indicates greater parent confidence.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 174 | 166
score on a scale
  baseline | 3.74 (0.72) | 3.73 (0.70)
  3-month follow up: number analyzed (Participants) | 160 | 161
  3-month follow up | 4.06 (0.57) | 3.78 (0.68)
  6-month follow up: number analyzed (Participants) | 155 | 154
  6-month follow up | 4.11 (0.61) | 3.78 (0.66)
  12-month follow up: number analyzed (Participants) | 155 | 153
  12-month follow up | 4.14 (0.57) | 3.91 (0.68)

5. Primary Outcome: Change From Baseline in Parent Alcohol Use
Description: Parent substance use was measured with the Opioid and Other Substance Use Involvement measure from the HEAL Prevention Cooperative Common Constructs. This measure assesses participants' use of alcohol, cannabis, prescription opioids, illegally manufactured opioids, and stimulants. A series of questions were asked about each substance of interest, starting with a question assessing if the parent had ever used the substance. Parents who responded "yes" received additional questions about that substance. Parents who responded "no" did not receive additional questions about that substance.
  Parents who indicated prior alcohol use were asked: "During the past 30 days, how many days did you drink alcohol?" Responses could range from 0-30 days. Higher scores indicate more frequent use of alcohol.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 169 | 162
days
  baseline | 2.88 (5.43) | 3.05 (5.22)
  3-month follow up: number analyzed (Participants) | 154 | 158
  3-month follow up | 2.38 (4.63) | 2.85 (4.98)
  6-month follow up: number analyzed (Participants) | 153 | 152
  6-month follow up | 2.43 (4.62) | 2.93 (5.61)
  12-month follow up: number analyzed (Participants) | 151 | 153
  12-month follow up | 1.88 (3.32) | 2.41 (4.37)

6. Primary Outcome: Change From Baseline in Parent Marijuana Use
Description: Parent substance use was measured with the Opioid and Other Substance Use Involvement measure from the HEAL Prevention Cooperative Common Constructs. This measure assesses participants' use of alcohol, cannabis, prescription opioids, illegally manufactured opioids, and stimulants. A series of questions were asked about each substance of interest, starting with a question assessing if the parent had ever used the substance. Parents who responded "yes" received additional questions about that substance; parents who responded "no" did not. The following header was included at the beginning of the section about marijuana use: "The next questions are about marijuana. Marijuana is also called pot, weed, or cannabis. These questions DO NOT include CBD only."
  Parents with prior marijuana use were asked: "During the past 30 days, how many days did you use marijuana?" Responses could range from 0-30 days. Higher scores indicate more frequent use of marijuana.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 133 | 137
days
  baseline | 4.58 (9.78) | 5.09 (9.98)
  3-month follow up: number analyzed (Participants) | 125 | 128
  3-month follow up | 5.02 (10.40) | 4.33 (9.38)
  6-month follow up: number analyzed (Participants) | 117 | 125
  6-month follow up | 4.32 (9.64) | 4.58 (9.52)
  12-month follow up: number analyzed (Participants) | 115 | 120
  12-month follow up | 4.43 (9.63) | 4.55 (9.71)

7. Primary Outcome: Change From Baseline in Parent Prescription Opioid Use
Description: Parent substance use was measured with the Opioid and Other Substance Use Involvement measure from the HEAL Prevention Cooperative. For each substance, parents were asked if they had ever used it. Parents who responded "yes" received additional questions; parents who responded "no" did not. A header in the section about use of prescription opioids read: "This next item asks about using prescription opioids for pain relief or treatment...in any way a doctor or medical provider did not tell you to use them. This includes:
  * Using without a prescription of your own (for example, someone else's medicine)
  * Using more or for longer than you were told to take it
  * Using for reasons other than pain (such as to get high, to sleep, or for anxiety)"
  Parents with prior prescription opioid misuse were asked: "During the past 30 days, how many days did you use a prescription opioid?" Responses could range from 0-30 days. Higher scores indicate more frequent use of prescription opioids.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 51 | 53
days
  baseline | 4.29 (10.38) | 4.98 (10.65)
  3-month follow up: number analyzed (Participants) | 42 | 43
  3-month follow up | 2.00 (6.95) | 3.37 (8.96)
  6-month follow up: number analyzed (Participants) | 40 | 41
  6-month follow up | 3.00 (9.12) | 4.59 (10.71)
  12-month follow up: number analyzed (Participants) | 36 | 40
  12-month follow up | 1.14 (5.06) | 2.30 (7.99)

8. Primary Outcome: Change From Baseline in Parent Use of Illegally Manufactured Opioids
Description: Parent substance use was measured with the Opioid and Other Substance Use Involvement measure from the HEAL Prevention Cooperative Common Constructs. This measure assesses participants' use of alcohol, cannabis, prescription opioids, illegally manufactured opioids, and stimulants. A series of questions were asked about each substance of interest, starting with a question assessing if the parent had ever used the substance. Parents who responded "yes" received additional questions about that substance; parents who responded "no" did not. The following header was included at the beginning of the section about illegally manufactured opioids: "The next questions ask about manufactured opioids including heroin (also called black tar, poppy, or smack) and Fentanyl."
  Parents with prior use of illegally manufactured opioids were asked: "During the past 30 days, how many days did you use heroin?" Responses could range from 0-30 days. Higher scores indicate more frequent use of heroin.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 24 | 26
days
  baseline | 1.25 (6.12) | 0.00 (0.00)
  3-month follow up: number analyzed (Participants) | 21 | 23
  3-month follow up | 1.43 (6.55) | 1.13 (5.42)
  6-month follow up: number analyzed (Participants) | 19 | 22
  6-month follow up | 0.21 (0.92) | 0.00 (0.00)
  12-month follow up: number analyzed (Participants) | 19 | 20
  12-month follow up | 1.11 (4.82) | 1.50 (6.71)

9. Primary Outcome: Change From Baseline in Parent Stimulant Use
Description: Parent substance use was measured with the Opioid and Other Substance Use Involvement measure from the HEAL Prevention Cooperative Common Constructs. A series of questions were asked about each substance of interest, starting with a question assessing if the parent had ever used the substance. Parents who responded "yes" received additional questions about that substance; parents who responded "no" did not. The following header was included at the beginning of the section about use of stimulants: "The next questions ask about stimulants. Some examples of stimulants include: Adderall, Concerta, Cylert, Provigil, Ritalin or Dexedrine, speed, amphetamine, methamphetamine, uppers, bennies, pep pills, crystal, crank."
  Parents with prior stimulant use were asked: "During the past 30 days, how many days did you use stimulants?" Responses could range from 0-30 days. Higher scores indicate more frequent use of stimulants.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 60 | 63
days
  baseline | 4.95 (10.48) | 5.70 (11.47)
  3-month follow up: number analyzed (Participants) | 51 | 54
  3-month follow up | 4.31 (10.09) | 3.48 (9.31)
  6-month follow up: number analyzed (Participants) | 48 | 49
  6-month follow up | 4.71 (10.50) | 4.18 (10.17)
  12-month follow up: number analyzed (Participants) | 46 | 46
  12-month follow up | 6.0 (11.42) | 2.57 (7.76)

10. Primary Outcome: Change From Baseline in Parental Depression
Description: Parental depression was measured with the Patient Health Questionnaire-9 (PHQ-9). Scores could range from 0-27; a higher score indicates greater depression.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning surveys at follow-up waves). Because no families were ever lost to follow-up or withdrew from the study, all families who participated at baseline were invited to participate at each follow-up wave. Thus, there are a few families who participated at 12-month follow-up who did not participate at an earlier follow-up wave.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 178 | 175
score on a scale
  Baseline | 8.14 (5.94) | 7.20 (5.74)
  3-month follow-up: number analyzed (Participants) | 168 | 169
  3-month follow-up | 6.38 (5.58) | 6.63 (5.45)
  6-month follow-up: number analyzed (Participants) | 161 | 164
  6-month follow-up | 6.17 (5.42) | 6.33 (5.50)
  12-month follow-up: number analyzed (Participants) | 164 | 161
  12-month follow-up | 6.10 (5.01) | 6.06 (5.02)

11. Primary Outcome: Change From Baseline in Parental Anxiety
Description: Parental anxiety was measured with the General Anxiety Disorder-7 (GAD-7). Scores could range from 0-21; a higher score indicates greater anxiety.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 177 | 175
score on a scale
  Baseline | 7.99 (5.73) | 7.41 (5.26)
  3-month follow up: number analyzed (Participants) | 168 | 169
  3-month follow up | 6.63 (5.31) | 6.90 (5.47)
  6-month follow up: number analyzed (Participants) | 160 | 164
  6-month follow up | 6.21 (5.31) | 6.54 (5.63)
  12-month follow-up: number analyzed (Participants) | 163 | 161
  12-month follow-up | 6.37 (5.27) | 6.03 (5.19)

12. Primary Outcome: Change From Baseline in Parental Stress
Description: Parental stress was measured with the Perceived Stress Scale. Scores could range from 0-56; a higher score indicates high perceived stress.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FCU Online + Coach | Waitlist Control
Number analyzed (Participants) | 178 | 175
score on a scale
  Baseline | 26.97 (8.80) | 26.60 (7.84)
  3-month follow up: number analyzed (Participants) | 167 | 169
  3-month follow up | 24.53 (8.38) | 25.56 (7.86)
  6-month follow up: number analyzed (Participants) | 162 | 164
  6-month follow up | 24.18 (8.62) | 25.37 (8.67)
  12-month follow up: number analyzed (Participants) | 165 | 160
  12-month follow up | 24.88 (8.16) | 25.15 (8.22)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the study period (until their 12-month post-test was completed).
Arm/Group | FCU Online + Coach | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/176
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/176
Other Adverse Events (participants affected / at risk) | 0/180 | 0/176

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT05180487/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT05180487/SAP_002.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT05180487/ICF_000.pdf